CLINICAL TRIAL: NCT03288337
Title: Impact of Hidradenitis Suppurativa on Quality of Life Functions: A Cross-Sectional Analysis of 400 Patients
Brief Title: Impact of Hidradenitis Suppurativa on Quality of Life Functions
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-3873
Record Dates: First submitted 2017-09-11; First posted 2017-09-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Hidradenitis Suppurativa; Quality of Life
Keywords: Hidradenitis Suppurativa; Quality of Life
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hidradenitis Suppurativa Cohort: Patients with HS who are eligible to fill out the series of quality of life questionnaires

SUMMARY:
The goal of this study is to get a better understanding of the impact of Hidradenitis Suppurativa (HS) on the quality of life of patients with this condition. Patients with HS will be asked questions about demographics including gender, age, and ethnicity. They will also be asked to complete questionnaires to determine how their skin condition affects their life. Study participation will last for 1 day, with potential for follow-up in the future. We hope this information will help us improve our treatment for this skin condition.

DETAILED DESCRIPTION:
The goal of this study is to get a better understanding of the impact of the skin condition, Hidradenitis Suppurativa, on quality of life function of patients. Patients with HS will be asked questions about demographics including gender, age, and ethnicity. They will also be asked to complete questionnaires to determine how their skin condition affects their life. The questionnaires include Beck Depression Inventory form, which gives us information how you feel about your skin condition and how it changes your mood; Dermatology Life Quality Index (DLQI), which gives us information about how your skin condition affects your quality of life; Skindex, which gives us more specific information about how your skin condition affects your quality of life; SF-36 health survey, which gives us information about your general health status; the Quality of Life Enjoyment and Satisfaction Questionnaire- short form (Q-LES-Q-SF), which gives us information on your enjoyment and satisfaction of your life; and the Employment/Productivity Health Economic Questionnaire, which will give us more information on your work and school status as well as household income. Study participation will last for 1 day, with potential for follow-up in the future. Through potential follow up visits we hope to determine the longitudinal effect of treatment modalities on QoL through future survey performance of the patient cohort. We hope this information will help us improve our treatment for this skin condition.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hidradenitis suppurativa
* Subject age >/= 18 years
* Able to be evaluated by a Montefiore physician

Exclusion Criteria:

* No clinical diagnosis of hidradenitis suppurativa
* Subject age < 18 years
* Subject unable to understand or answer provided questionnaires
* Unable to evaluated by a Montefiore physician

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy adults (ages 18-99) who have a diagnosis of HS (as deemed by a physician at the Hidradenitis Suppurativa Treatment Center at Montefiore Medical Center)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Dermatology-related quality of life | Baseline
  Quality of life as measured using standardized Dermatology Quality of Life Index
Presence and severity of depression | Baseline
  Presence and severity of depression as measured using standardized Beck Depression Inventory
Dermatology-related quality of life | Baseline
  Quality of life as measured using standardized SkinDex questionnaires
Subject-reported subject health | Baseline
  Subject-reported subject health as measured using standardized SF-36 questionnaires
Degree of enjoyment and satisfaction experienced by subjects in daily functioning. | Baseline
  Degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning as measured by the standardized Quality of Life Enjoyment and Satisfaction Questionnaire-short form.
Employment and economic productivity | Baseline
  Self-reported employment and economic productivity as measured by a standardized health economic questionnaire

SECONDARY OUTCOMES:
Change in quality of life | At 6 months
  Change in quality of life as measured using standardized Dermatology Quality of Life Index after treatment initiation
Change in presence and severity of depression as measured using standardized Beck Depression Inventory | At 6 months
  Change in presence and severity of depression as measured using standardized Beck Depression Inventory after treatment initiation
Change in quality of life | At 6 months
  Change in quality of life as measured using standardized SkinDex questionnaires after treatment initiation
Change in subject-reported subject health | At 6 months
  Change in subject-reported subject health as measured using standardized SF-36 questionnaires after treatment initiation
Change in degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning | At 6 months
  Change in degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning as measured by the standardized Quality of Life Enjoyment and Satisfaction Questionnaire-short form after treatment initiation
Change in self-reported employment and economic productivity | At 6 months
  Change in self-reported employment and economic productivity as measured by a standardized health economic questionnaire after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cohen, MD. MPH, Principal Investigator — Momtefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data to other researchers

REFERENCES:
- See also: Montefiore Hidradenitis Suppurativa Website — http://www.montefiore.org/hidradenitis-suppurativa